CLINICAL TRIAL: NCT04328272
Title: Effectiveness of Hydroxychloroquine in Covid-19 Patients: A Single Centred Single-blind RCT Study
Brief Title: Effectiveness of Hydroxychloroquine in Covid-19 Patients
Acronym: Covid
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Dr. Umar Farooq (Other)
Collaborators: Ayub Medical College, Abbottabad (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Umar Farooq, Dean & Chief Executive Officer, Ayub Medical College, Abbottabad
Organization: Ayub Medical College, Abbottabad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ath/ct101/22/3
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: COVID19
Keywords: covid 19; treatment
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin; Glucose; Aspartame

STUDY DESIGN:
Intervention Model Description: three parallel groups randomly asserted for intervention
Who Masked: Participant
Masking Description: Single blinded:
  As, the disease is novel and putting the lives at risk is unethical. therefore, It is important for investigator to know the group and carry close regular monitoring of participants so that proper further intervention can be made when required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydroxychloroquine (Experimental): tablet hydroxychloroquine (HCQ). Day-1 (initial) 1st dose, 3 tablets (200 mg per tablet), 2nd dose after 6 hours, 3 tablets (200 mg per tablet) per oral. From day 2 to 7 (maintenance dose), 2 tablets twice a day.
  Interventions: Drug: Hydroxychloroquine 200 Mg Oral Tablet
- Azithromycin (Active Comparator): Tablet azithromycin (AZC) 500 mg orally as a single dose on day 1, followed by 250 mg orally once a day on days 2 to 7.
  Interventions: Drug: Hydroxychloroquine 200 Mg Oral Tablet; Drug: Azithromycin 500Mg Oral Tablet
- Suger Tablets (Placebo Comparator): Placebo (sugar tablet) twice daily for 7 days
  Interventions: Dietary Supplement: Glucose tablets

INTERVENTIONS:
Drug: Hydroxychloroquine 200 Mg Oral Tablet — Hydroxychloroquine administered orally with water
  Other Names: Plaquenil
  Arms: Azithromycin; Hydroxychloroquine
Drug: Azithromycin 500Mg Oral Tablet — Azithromycin administered orally with water
  Other Names: Zetro
  Arms: Azithromycin
Dietary Supplement: Glucose tablets — administered orally with water
  Other Names: Canderel
  Arms: Suger Tablets

SUMMARY:
To find the effectiveness of hydroxychloroquine alone and adjuvant with azithromycin in mild to severe Covide-19 pneumonia patients admitted to Coronavirus cell/ward of Ayub Teaching hospital, Abbottabad Pakistan. A single centered, single-blind randomized control trial study.

DETAILED DESCRIPTION:
Coronavirus (SARS-nCoV-2) is a member family coronaviridae, order Nidovirales. It is single-stranded, positive sense enveloped RNA discovered in early 1960s. Coronavirus pandemic put a lot of lives at stake. By 19 March 2020, a total of 219238 confirmed cases with 8967 being dead and 85742 recovered cases have been reported. Worldwide, in 9 days, the confirmed death cases have been doubled. The average death rate of Covid-19 per day is approximately 88 patients as of the given date. Unlike, SARS-CoV and MERS-CoV, the disease progression and mortality rate of Covid-19 is startling. The pre-pathogenic course of novel Covid-19 is yet to be determined, so the risk factors, clinical picture and medical intervention too. Only supportive therapy is being practised. Yet many trials of antimalarial drug, chloroquine and quinolone is currently taking place worldwide. According to Cortegiani A, 23 ongoing trials from China have been registered. Clinical experience from recent Wuhan epidemic came up with promising results of chloroquine and hydroxychloroquine in Covid-19 positive patients. Some in-vitro studies suggest that these immunomodulant drugs can interfere with SARS-nCov-2 replication. These are federal drug authority approved medicine for malaria. Yet their effectiveness and safety in treating Covid-19 pneumonia is a question mark.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases of Covid-19 (all by RT-PCR from same laboratory)
* Mild to severe clinical presentation (identified at the time of admission to ward by National Early Warning Score NEWS-2; mild 0-4; severe 5-6)

Exclusion Criteria:

* Covid-19 critically ill patients (NEWS-2 score <7),
* Unable to take oral medication,
* Immunocompromised,
* Creatinine clearance (CCL) < 30 ml/min,
* Aspartate transaminase (AST) or alanine transaminase (ALT) > 5 times Upper limit of normal (ULN),
* d-dimer > 2microgram per liter, or
* Known comorbid condition like hypertension, cardiovascular disease, diabetes mellites, asthma, COPD, cerebrovascular disorder, malignancy of any type, pregnancy,
* BMI less than 18
* Smoking history (one pack per day) for past six months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-03-28 (Estimated); Primary Completion 2020-05-28 (Estimated); Study Completion 2020-06-28 (Estimated)

PRIMARY OUTCOMES:
National Early Warning Score equal to zero | 3-5 Days
  National Early Warning Score equal to zero is when patients recovered clinically. Respiration 14-20breaths/minute, oxygen saturation percent greater than 96, (without breathing aid), systolic blood pressure 111-180 mmhg, pulse 60-90 beats.minute, alert consciousness and 35.1-38 degree Celsius body temperature.

SECONDARY OUTCOMES:
C-reactive proteins | 3-5 Days
  below 3.0 miligram/Liter of blood sample
Lymphocyte Count | 3-5days
  1000 -4800 lymphocytes in 1 microliter of blood
d-dimers | 3-5days
  less than 250 ng/mL, or less than 0.4 mcg/mL of blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Umar Farooq, PhD, Principal Investigator — Khyber Medical University Peshawer
Locations (1):
- Ayub Teaching Institution, Abbottābād, K.p.k, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
as each individual will have his/her own coded file. the required data from each will be extracted and will be made available in soft copies